CLINICAL TRIAL: NCT01399632
Title: Dietary Fat and High-Density Lipoprotein (HDL) Metabolism-Effect of Carbohydrate and Fat Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Frank M. Sacks, MD, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: HL095964
Record Dates: First submitted 2011-07-15; First posted 2011-07-22 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Overweight; Cardiovascular Diseases
MeSH Terms: conditions — Overweight; Cardiovascular Diseases | interventions — Diet, Fat-Restricted; Diet; Diet, Carbohydrate-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Fat and Low Carbohydrate Diet (Experimental)
  Interventions: Behavioral: High Fat and Low Carbohydrate Diet
- Low Fat and High Carbohydrate Diet (Experimental)
  Interventions: Behavioral: Low Fat and High Carbohydrate Diet

INTERVENTIONS:
Behavioral: Low Fat and High Carbohydrate Diet — Low Fat and High Carbohydrate Diet
  Other Names: Diet and HDL Metabolism
  Arms: Low Fat and High Carbohydrate Diet
Behavioral: High Fat and Low Carbohydrate Diet — High Fat and Low Carbohydrate Diet
  Other Names: Diet and HDL Metabolism
  Arms: High Fat and Low Carbohydrate Diet

SUMMARY:
Generally, people with low levels of high-density lipoprotein (HDL) in blood are more likely to get heart disease than those who have normal or high levels. Dietary fat, whether the harmful type (saturated) or beneficial type (unsaturated) raises HDL levels. Dietary carbohydrate lowers HDL. The investigators are doing this research study to find out why the amount of HDL in a person's blood is affected by dietary unsaturated fat and carbohydrate. The investigators will trace the ability of the HDL in a person's blood to take up cholesterol, get bigger, and then leave the blood by passing into the liver. The investigators want to know if dietary unsaturated fat improves the ability of HDL to do this compared to dietary carbohydrate.

DETAILED DESCRIPTION:
The investigators will study the kinetics of multiple types of high-density lipoprotein (HDL) in humans under two strictly controlled dietary conditions, high unsaturated fat and high carbohydrate, in 20 individuals with low HDL cholesterol and overweight or obesity. The participants will be given the controlled diets for 4 weeks in a randomized crossover design. They will be admitted to the Brigham & Women's Hospital Center for Clinical Investigation (CCI) the morning of Day 28 when they will be infused intravenously with a stable isotope tracer, trideuterated (D3), leucine for 10 minutes as a bolus. Blood will be sampled in the hospital through 24 hours, and thereafter at the ambulatory clinical center throughout 94 hours. HDL subtypes will be prepared in Dr. Sacks's laboratory at Harvard School of Public Health (HSPH) and analyzed for content of lipids and proteins, and for incorporation of the tracer into apolipoprotein A-I, the principal protein of HDL. These data will be studied by interactive modeling to a multi-compartment model of human HDL physiology that best fits the observed data. The model will yield HDL metabolic rates during unsaturated fat and carbohydrate-rich diets which will be tested for statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Only accepting participants in the Boston, Massachusetts area
* Age 21 to 75, male or female
* Willingness to eat prescribed diet for 4 weeks prior to infusion date, and 3.5 days after the infusion date
* Willingness to participate in an infusion protocol, which will require them to stay at the Center for Clinical Investigation (CCI) for one night and return for blood draws every day for the next 3 days.
* Body Mass Index (BMI) 25-35 Kg/m2
* HDL<45 mg/dL for men, <55 mg/dL for women

Exclusion Criteria:

* Hematocrit <33
* Low-density Lipoprotein (LDL) cholesterol >190 mg/dl
* HDL cholesterol <20 mg/dl, to exclude those with rare genetic HDL deficiency syndromes
* Fasting Triglycerides >500 mg/dl to exclude those with risk of pancreatitis
* ApoE genotypes, E2E2, E2E4, and E4E4.
* Lipid lowering medications
* Hormone replacement therapy
* Other medicines that affect plasma lipid levels: e.g. beta blockers, certain psychiatric medicines including Alprazolam, Chlordiazepoxide, Clonazepam, Diazepam, Lorazepam, Oxazepam, Prazepam, Aripiprazole, Chlorpromazine, Chlorprothixene, Clozapine, Flupenthixol, Fluphenazine, Haloperidol, Loxapine, Mesoridazine, Methotrimeprazine, Molindone, Olanzapine, Perphenazine, Pimozide, Pipotiazine, Prochlorperazine, Promazine, Promethazine, Quetiapine, Risperidone, Sulpiride, Thioridazine, Thiothixene, Trifluoperazine, Ziprasidone.
* Thyrotrophin-stimulating hormone: <0.5 or >5.0
* alanine aminotransferase : 1.5 x uln or 60 IU/L
* Aspartate transaminase: 1.5 x uln or 60 IU/L
* Bilirubin: outside upper limit. (>1.2 mg/dL)
* Creatinine: outside upper limit (>1.00 mg/dL)
* Diabetes by history
* Diabetes by fasting or post-challenge glycemia according to ADA guidelines:

  * Fasting hyperglycemia (glucose >126 mg/dl).
  * Post-challenge glucose by standard oral glucose tolerance test, >200 mg/dl
* Will not eat the provided diet and abstain from alcoholic beverages.
* Women who are pregnant

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
high-density lipoprotein (HDL) cholesterol | Diet Periods I and II-Days 28-32
  To determine how dietary unsaturated fat when it replaces carbohydrate affects HDL metabolism.

SECONDARY OUTCOMES:
To study HDL with apoE | Diet Periods I and II-Days 28-32

OTHER OUTCOMES:
Provide guidance for interpreting effects of unsaturated fats on reverse cholesterol transport | Diet Periods I and II-Days 28-32

CONTACTS AND LOCATIONS:
Overall Officials: Frank M Sacks, MD, Principal Investigator — Harvard University
Locations (1):
- Harvard T. H. Chan School of Public Health, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Morton AM, Furtado JD, Mendivil CO, Sacks FM. Dietary unsaturated fat increases HDL metabolic pathways involving apoE favorable to reverse cholesterol transport. JCI Insight. 2019 Apr 4;4(7):e124620. doi: 10.1172/jci.insight.124620. eCollection 2019 Apr 4. PMID 30944249
- [Derived] Morton AM, Koch M, Mendivil CO, Furtado JD, Tjonneland A, Overvad K, Wang L, Jensen MK, Sacks FM. Apolipoproteins E and CIII interact to regulate HDL metabolism and coronary heart disease risk. JCI Insight. 2018 Feb 22;3(4):e98045. doi: 10.1172/jci.insight.98045. eCollection 2018 Feb 22. PMID 29467335